CLINICAL TRIAL: NCT02870127
Title: Genetic Study of Varicose Disease by Sequencing Exome
Brief Title: Clinical Investigation and Molecular Forms of Family Disease of Varicose
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC12_0142
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples and venous tissues of patients
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: blood sample

SUMMARY:
The existence of a family factor in the genesis of varicose veins is certain, but few studies have addressed reliably instead of the genetic factor in clinical and molecular level. The investigator initiated an original study to identify one or more genetic abnormalities predisposing to varicose disease, based on a combined approach of genetic linkage and of exome sequencing. The clinical research phase is an essential prerequisite to the identification of genetic mutations; it is to identify large affected families and ensure an extremely rigorous and accurate phenotyping of individuals over several generations. A first clinical work has identified and / or phenotype 8 families with a genetically informative family suggesting autosomal dominant inheritance. Linkage analysis suggested several candidate chromosomal regions without allowing the identification of a gene. This project aims to resume and expand the Family clinical investigations and apply the techniques of genome analysis points, including exome sequencing on the most informative families to identify the genes and mechanisms responsible of this disease and improve the prevention and the treatment of varicose veins.

ELIGIBILITY:
Inclusion Criteria:

* Any patient consultant the Medicine Vascular Surgery for varicose veins of the lower limbs as part of a manifesto family context
* Varices Presence in at least one family member
* Written consent

Exclusion Criteria:

* Patients who are unable to sign or who refuse to sign an informed consent
* Subjects aged less than 25 years, due to the low penetrance of varicose disease that age.
* Secondary veins at a post-thrombotic disease (suspected by the examination and confirmed by Doppler ultrasonography of the deep venous system)
* Venous angiodysplasia or secondary varicose arteriovenous fistulas.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The initial step of this protocol relies on recruiting large families (> 8 met) for a genetic linkage analysis. It consists firstly in identifying patients with varicose veins occurring in a family context, and to conduct a comprehensive survey to assess the potentially informative family (significant number of individuals with multiple generations) and ensure their membership prior to the study. The next step is the fine and accurate phenotyping of each of the family members and the collection of a blood sample for DNA extraction for molecular genetic analysis (family linkage analysis and sequencing exome ).
Sampling Method: Non-Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2016-12-19 (Actual)

PRIMARY OUTCOMES:
genetic abnormalities segregating with the presence of varicose veins in the informative families recruited. | year 4

SECONDARY OUTCOMES:
genotype/phenotype relationship | year 4
  improving knowledge of the genotype / phenotype based on genes identified in different families.

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Antoine Pistorius, PU-PH, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - La Roche sur Yon Hospital, La Roche-sur-Yon
  - Nantes Univesrity Hospital, Nantes

IPD SHARING:
Plan to Share IPD: Undecided